CLINICAL TRIAL: NCT01128959
Title: Open-Label Study to Assess the Safety and Tolerability of Intravenous Carbamazepine as Short-Term Replacement of Oral Carbamazepine in Adult Patients With Epilepsy
Brief Title: Study to Assess the Safety and Tolerability of Intravenous Carbamazepine in Adults With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lundbeck LLC (Industry)
Collaborators: Ligand Pharmaceuticals (Industry); ICON Clinical Research (Industry); Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13181A
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Epilepsy
Keywords: Epilepsy; Intravenous Carbamazepine; Oral Carbamazepine
MeSH Terms: conditions — Epilepsy | interventions — Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous Carbamazepine (IV CBZ) (Experimental)
  Interventions: Drug: Intravenous Carbamazepine (IV CBZ)

INTERVENTIONS:
Drug: Intravenous Carbamazepine (IV CBZ) — 10 mg/mL of IV CBZ dissolved in 250 mg/mL of Captisol® (sulfobutylether-beta-cyclodextrin) dosed at 70% of the patient's daily maintenance dose of oral CBZ administered after suitable dilution with D5W by IV infusion every 6 hours.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of intravenous (IV) carbamazepine (CBZ) administered as multiple 15 minute infusions and a single 5 minute infusion to adult patients with epilepsy on stable higher doses of oral CBZ.

DETAILED DESCRIPTION:
This was a phase III, multicenter, open-label study designed to assess the safety and tolerability of intravenously administered CBZ in adult patients with epilepsy. This study included a 28 day Lead-in Period, a Confinement Period (up to 7 days and 6 nights) and a 28 day Follow-up Period.

Patients began confinement on Day -1 of the trial, continuing to take their oral CBZ as prescribed by the investigator. On the morning of Day 0, Day 4, and Day 17, patients began the 24hr urine collection for evaluation of urinary biomarkers. All patients temporarily discontinued their prescribed oral CBZ and begin IV CBZ administration on the morning of Day 1, continuing administrations every 6 hours (Q6h) through the morning of Day 4.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or legal representative must be able to read, understand, sign and date the IRB approved Informed Consent Form and HIPAA Authorization prior to study participation.
2. The patient is a man or a non-pregnant woman who is at least 18 years of age.
3. If a woman:

   * Patient is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomay or hysterectomy), or if childbearing potential, must comply with a method of birth control acceptable to the investigator during the study, for at least 28 days prior to Day 1 and for 28 days following completion of the study.
   * Patient is not breastfeeding.
   * Patient of childbearing potential must have a negative serum pregnancy test at Day -28 and a negative urine pregnancy test or serum pregnancy test at Day -1.
4. The patient is diagnosed with any of the approved epilepsy indications for CBZ:

   * Partial seizures with complex symptomatology (psychomotor, temporal lobe)
   * Generalised tonic clonic seizures (GTCS) (grand mal): myoclonic, clonic, tonic, tonic-clonic, atonic
   * Mixed seizure patterns that include the above, or other partial or generalised seizures (except absence seizures - please see exclusion point number 12)
5. The patient is receiving a stable dose of oral CBZ (tablet or capsule formulation) of 1200 mg/day to 2000 mg/day, for a minimum of 14 days prior to Day -28.
6. The patient is receiving a constant dose of all other concomitant medications used for chronic conditions, (including OTC medications and herbal supplements) for a minimum of 28 days prior to Day 1.
7. The patient is not expected to have any change in his/her baseline AED treatment during the treatment period.
8. The patient is able to comply with maintaining an accurate Seizure and antiepileptic drug diary.
9. The patient is able to comply with all study procedures including complying with protocol determined dosing intervals, confinement at the investigative site for up to 6 nights and 7 days, and agrees to participate in the entire study.

Exclusion Criteria:

1. The patient has a known hypersensitivity to CBZ, Captisol, or to any of the tricyclic compounds, such as amitriptyline, trimipramine, imipramine; oxacarbazepine, phenytoin, or their analogues or metabolites.
2. The patient has a history of previous bone marrow depression.
3. The patient has a history of intolerance to IV administration of medication.
4. The patient is pregnant or lactating.
5. The patient is being treated with a monoamine oxidase (MAO) inhibitor.
6. The patient is using oral, intramuscular, or any other hormone delivery method as their primary form of birth control.
7. The patient has an ECG with corrected QT interval by Fridericia's correction formula (QTcF) greater than 450 msec at Screening or Day -1.
8. The patient has a screening ALT, AST or bilirubin >=3 times the upper limit of normal.
9. The patient has an estimated ClCR (based of Cockcroft-Gault) of <50 ml/min.
10. The patient has had a clinically significant illness/infection or has had any surgical procedure within 30 days prior to Screening.
11. The patient has a significant history of cardiac, renal, neurologic (other than epilepsy), psychiatric, oncologic, endocrinologic, metabolic, or hepatic disease, which would adversely affect their participation in this study.
12. The patient is receiving oral CBZ for absence seizures.
13. The patient has had an episode of status epilepticus within 4 weeks of Screening.
14. The patient has a history of severe or serious adverse reactions to CBZ (for example, aplastic anemia, agranulocytosis, SJS.
15. The patient has taken or used any investigational drug or device in the 30 days prior to Screening.
16. The patient has previously been administered IV CBZ in a previous clinical trial (for example OV-1015).
17. The patient has a urine toxicology screen positive for phencyclidine, benzodiazepines (unless due to the patient's concomitant AEDs), cannabinoids, cocaine, amphetamines, opiates, barbiturates (unless due to the patient's concomitant AEDs), or alcohol at Screening or Day -1.
18. The patient has had a diagnosis of drug or alcohol abuse within the past year prior to Screening.
19. The patient has had significant blood loss (>500 mL) or donation within 14 days of Screening.
20. The patient has a history of poor oral CBZ compliance.
21. The patient is participating in a weight loss or nicotine cessation program.
22. The patient has a history of increased intraocular pressure or is on medication for glaucoma.
23. The patient is considered by the investigator to be an unsuitable candidate for the study, which may include an increase in the frequency, severity and duration of seizures during the Pre-Treatment Period (Days -28-0).
24. The patient has previously participated in this study.
25. The patient is a member of the site personnel or their immediate families.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (29):
- United States (29):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Clinical Trials Incorporated, Little Rock, Arkansas
  - Collaborative Neuroscience Network, Inc., Torrance, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - University of South Florida, Tampa, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Southern illinois University School of Medicine, Springfield, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Via Christi Epilepsy Center, Wichita, Kansas
  - Leonard J. Chabert Medical Center, Houma, Louisiana
  - Louisiana Research Associates, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota & Prism Research, Saint Paul, Minnesota
  - The Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - Langone Medical Center NYU Comprehensive Epilepsy Center, New York, New York
  - Columbia University Medical Center: Dept of Neurology, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medicical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University Health systems, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Neurological Clinic of Texas, P.A., Dallas, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - University of Virginia, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia

REFERENCES:
- [Derived] Lee D, Kalu U, Halford JJ, Biton V, Cloyd J, Klein P, Bekersky I, Peng G, Dheerendra S, Tolbert D. Intravenous carbamazepine as short-term replacement therapy for oral carbamazepine in adults with epilepsy: Pooled tolerability results from two open-label trials. Epilepsia. 2015 Jun;56(6):906-14. doi: 10.1111/epi.12991. Epub 2015 Apr 25. PMID 25912051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited through physician referrals and/or recruitment methods at hospitals and clinics. Advertisements were used by 5 sites.
Period: Lead in Period
Arm/Group | Intravenous Carbamazepine (IV CBZ)
Started | 108
Completed | 105
Not Completed | 3
Not completed — Adverse Event | 3
Period: Treatment Period
Arm/Group | Intravenous Carbamazepine (IV CBZ)
Started | 105
Completed | 101
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous Carbamazepine (IV CBZ)
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 72
  More than one race | 0
  Unknown or Not Reported | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 86
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Time Frame: Baseline to after last iv dose on day 4
Population: All Patients Treated Set
Measure: Number; unit: Number of adverse events
Groups:
- Intravenous Carbamazepine (IV CBZ) 15 Minutes Infusion; Intravenous Carbamazepine (IV CBZ) 5 Minutes Infusion: Intravenous Carbamazepine (IV CBZ): 10 mg/mL of IV CBZ dissolved in 250 mg/mL of Captisol® (sulfobutylether-beta-cyclodextrin) dosed at 70% of the patient's daily maintenance dose of oral CBZ administered after suitable dilution with D5W by IV infusion every 6 hours.
Arm/Group | Intravenous Carbamazepine (IV CBZ) 15 Minutes Infusion | Intravenous Carbamazepine (IV CBZ) 5 Minutes Infusion
Number analyzed (Participants) | 105 | 101
Number of adverse events | 126 | 26

ADVERSE EVENTS:
Time Frame: Baseline to to after last iv dose on day 4
Arm/Group | Intravenous Carbamazepine (IV CBZ) 15 Minutes Infusion | Intravenous Carbamazepine (IV CBZ) 5 Minutes Infusion
Serious Adverse Events (participants affected / at risk) | 2/105 | 0/101
Other Adverse Events (participants affected / at risk) | 29/105 | 11/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Carbamazepine (IV CBZ) 15 Minutes Infusion (N=105) | Intravenous Carbamazepine (IV CBZ) 5 Minutes Infusion (N=101)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Carbamazepine (IV CBZ) 15 Minutes Infusion (N=105) | Intravenous Carbamazepine (IV CBZ) 5 Minutes Infusion (N=101)
Dizziness (Nervous system disorders) | 20 | 11
Headache (Nervous system disorders) | 9 | 0
Somnolence (Nervous system disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No